CLINICAL TRIAL: NCT00770497
Title: Effect of Pioglitazone Compared to a Combination Therapy With Ramipril and to a Ramipril Monotherapy on Low Grade Inflammation and Vascular Function in Patients With Increased Cardiovascular Risk and an Activated Inflammation. A Randomized Double-blinded Phase II Study.
Brief Title: Efficacy Study of Pioglitazone and Ramipril Combination Therapy in Treating Non-diabetic Hypertensive Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Pharma GmbH, Aachen (Germany)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATS K023; 2006-004028-35 (EudraCT Number); D-PIO-110 (Other: Takeda ID); U1111-1115-9194 (Registry Identifier: WHO); NCT00975624 (obsolete NCT alias)
Record Dates: First submitted 2008-10-09; First posted 2008-10-10 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Inflammation; Hypertension
Keywords: drug effects; Hypertension; Vascular Resistance; Drug Therapy; physiopathology, vascular
MeSH Terms: conditions — Inflammation; Hypertension | interventions — Pioglitazone; Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pioglitazone 15 mg to 30 mg QD (Experimental)
  Interventions: Drug: Pioglitazone
- Pioglitazone 15 mg to 30 mg QD + Ramipril 2.5 mg to 5 mg QD (Active Comparator)
  Interventions: Drug: Pioglitazone and ramipril
- Ramipril 2.5 mg to 5 mg QD (Active Comparator)
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 15 mg, tablets, orally, once daily and ramipril placebo-matching tablets, orally, once daily for two weeks; increased to:
  Pioglitazone 30 mg, tablets, orally, once daily and ramipril placebo-matching tablets, orally, once daily for up to 10 weeks.
  Other Names: ACTOS®; AD4833
  Arms: Pioglitazone 15 mg to 30 mg QD
Drug: Pioglitazone and ramipril — Pioglitazone 15 mg, tablets, orally, once daily and ramipril 2.5 mg, tablets, orally, once daily for two weeks; increased to:
  Pioglitazone 30 mg, tablets, orally, once daily and ramipril 5 mg, tablets, orally, once daily for up to 10 weeks.
  Other Names: ACTOS®; AD4833
  Arms: Pioglitazone 15 mg to 30 mg QD + Ramipril 2.5 mg to 5 mg QD
Drug: Ramipril — Pioglitazone placebo-matching tablets, orally, once daily and ramipril 2.5 mg, tablets, orally, once daily for two weeks; increased to:
  Pioglitazone placebo-matching tablets, orally, once daily and ramipril 5 mg, tablets, orally, once daily for up to 10 weeks.
  Arms: Ramipril 2.5 mg to 5 mg QD

SUMMARY:
The purpose of this study is to determine the effects of pioglitazone, once daily (QD), on low grade inflammation and vascular function in hypertensive patients.

DETAILED DESCRIPTION:
Patients with insulin resistance and an activated inflammation are prone for cardiovascular complications like myocardial infarction or stroke. Pharmacological interventions reducing vascular inflammation are thought to reduce cardiovascular risk in diabetic and in non-diabetic patients.

Intervention with ACE inhibitors like ramipril is an established and widely used treatment for patients with high blood pressure, proven to reduce cardiovascular risk. Treatment of non-diabetic patients with pioglitazone has shown to improve the cardiovascular risk profile in non-diabetic patients beyond its effect on blood glucose levels.

The purpose of this study is to evaluate effects on low grade inflammation and vascular function of pioglitazone in non-diabetic, hypertensive patients with pre treatment with angiotensin converting enzyme inhibitors (that will be replaced by the study medication at time of randomization).

ELIGIBILITY:
Inclusion Criteria:

* Has arterial hypertension.
* Is on stable treatment with an Angiotensin Converting Enzyme inhibitor at least for 12 weeks.
* Has a high sensitive C-Reactive Protein value greater than 1.0 mg/L and less than 10.0 mg/L.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* Manifests or has newly detected diabetes mellitus type 2 according to World Health Organization criteria.
* Has Type 1 Diabetes.
* Has acute infections.
* Chronic inflammatory diseases which cause elevated CRP-values (e.g. rheumatic diseases, pyelonephritis or osteomyelitis).
* Use of acetyl salicylic acid and/or Non-steroidal Anti-inflammatory Drugs or Cox-2-inhibitors within the last 4 weeks prior to screening visit, use of Rifampicin within the last 12 weeks prior to screening visit.
* Uncontrolled hypertension (repeated blood pressure greater than 180/100 mmHg for at least three times within two weeks); persistent hypotension (systolic less than 90 mmHg) or hemodynamic instability.
* Anamnestic history of hypersensitivity to the study drugs or to drugs with similar chemical structures.
* History of severe or multiple allergies.
* Treatment with any other investigational drug within 3 months before trial entry.
* Has a progressive, fatal disease.
* History of drug or alcohol abuse within the last 5 years.
* A history of significant cardiovascular (New York Heart Association stage I - IV, hemodynamic relevant aortic or mitral valve stenosis, hypertrophic obstructive cardiomyopathy), respiratory, gastrointestinal, hepatic (alanine aminotransferase greater than 2.5 times the normal reference range), renal (creatinine greater than 2.0 mg/dL), or hematological disease, history of macular edema.
* State after kidney transplantation, hemodynamic relevant renal artery stenosis (bilateral or unilateral in case of single kidney).
* Blood donation within the last 30 days.
* Serum potassium greater than 5.5 mmol/L.
* History of hyperaldosteronism.
* Treatment with thiazolidinediones within 3 months prior to screening.
* Acute myocardial infarction, open heart surgery or cerebral events (stroke/transient ischemic attack) within 30 days prior to screening visit.
* If statin therapy applicable: Change of medication within the last 12 weeks.
* History of angioneurotic edema (hereditary or idiopathic as consequence of previous Angiotensin Converting Enzyme inhibitor treatment).
* Dialysis or hemofiltration.
* Low Density Lipoprotein apheresis with dextran sulphate.
* Allergic to toxic agents derived from insects.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Change in the high-sensitivity C-reactive Protein value. | Week: 12.

SECONDARY OUTCOMES:
Change from Baseline in Glucose tolerance as assessed by an oral glucose tolerance test. | Week: 12.
Change from Baseline in Insulin sensitivity according to the Homeostatic Model Assessment - Sensitivity score and Insulin Secretion. | Weeks: 6 and 12.
Change from Baseline in Glycosylated Hemoglobin levels. | Week: 12.
Change from Baseline in C-Peptide levels. | Weeks: 6 and 12.
Change from Baseline in Proinsulin intact levels. | Weeks: 6 and 12.
Change from Baseline in 24 hours Blood Pressure Profile. | Week: 12.
Change from Baseline in high-sensitivity C-reactive Protein levels. | Weeks: 6 and 10.
Change from Baseline in Adiponectin levels. | Weeks: 6 and 12.
Change from Baseline in Monocyte Chemoattractant Protein-1 levels. | Weeks: 6 and 12.
Change from Baseline in Matrix metalloproteinase-9 levels. | Weeks: 6 and 12.
Change from Baseline in P-selectin levels. | Weeks: 6 and 12.
Change from Baseline in Plasminogen Activator Inhibitor-1 levels. | Weeks: 6 and 12.
Change from Baseline in Relaxin levels. | Weeks: 6 and 12.
Change from Baseline in Endothelin 1-21 levels. | Weeks: 6 and 12.
Change from Baseline in Nitrotyrosine levels. | Weeks: 6 and 12.
Change from Baseline in Asymmetric Dimethylarginine levels. | Weeks: 6 and 12.
Change from Baseline in Myeloperoxidase levels. | Weeks: 6 and 12.
Change from Baseline in levels of Oxidative Stress as assessed by Per-Ox-Assay. | Weeks: 6 and 12.
Change from Baseline in Total Cholesterol levels. | Weeks: 6 and 12.
Change from Baseline in Triglycerides levels. | Weeks: 6 and 12.
Change from Baseline in High Density Lipoprotein levels. | Weeks: 6 and 12.
Change from Baseline in Low Density Lipoprotein levels. | Weeks: 6 and 12.
Change from Baseline in Oxidized Low Density Lipoprotein levels. | Weeks: 6 and 12.
Change from Baseline in Soluble Intercellular Adhesion Molecule levels. | Weeks: 6 and 12.
Change from Baseline in Soluble Vascular Cell Adhesion Molecule levels. | Weeks: 6 and 12.
Change from Baseline in Osteoprotegrin levels. | Weeks: 6 and 12.
Change from Baseline in 11-dihydroxy-thromboxan B2 levels. | Weeks: 6 and 12.
Change from Baseline in Placental Growth Factor levels. | Weeks: 6 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Adviser Clinical Research, Study Director — Takeda Pharma Gmbh, Aachen (Germany)
Locations (13):
- Germany (13):
  - Deggingen, Baden-Wurttemberg
  - Rottweil, Baden-Wurttemberg
  - Spaichingen, Baden-Wurttemberg
  - Weilersbach, Bavaria
  - Hanover, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Werne, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Schauenburg, Rhineland-Palatinate
  - Dresden, Saxony
  - Berlin, State of Berlin
  - Blankenhain, Thuringia

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI